CLINICAL TRIAL: NCT03395288
Title: Randomized, Controlled Trial to Determine the Efficacy of Nutraceutical vs Control as Non-antibiotic Prophylaxis for Recurrent Urinary Tract Infection in Postmenopausal Women Using Vaginal Estrogen Therapy
Brief Title: Nutraceutical Efficacy for rUTI
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Performed a futility analysis and determined that study objectives could not be met.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201711120
Record Dates: First submitted 2017-12-28; First posted 2018-01-10 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Urinary Tract Infections
Keywords: UTI; recurrent UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Mannose

STUDY DESIGN:
Intervention Model Description: There will be a RCT portion of the study with a treatment arm and a control arm and an additional observational arm of the study.
Who Masked: Participant
Masking Description: Participants in the RCT treatment and RCT control arm will not be told the name of the nutraceutical being studied. Participants in the observational arm will be aware of the nutraceutical being studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RCT treatment arm (Experimental): Participants in this arm will dissolve one (1) level teaspoon of the nutraceutical powder (D-mannose) in at least 200 ml of water one time a day, approximately every 24 hours. (200 ml of water = 6.7 fluid ounces). Duration of study drug is 90 days.
  Interventions: Drug: D-Mannose
- RCT control arm (No Intervention): Participants in this arm will not use any additional intervention.
- Observational arm (Experimental): Participants in this arm will either take a total of 1000 mg D-mannose in capsule form every 12 hours OR they will dissolve one (1) level teaspoon of the nutraceutical powder (D-mannose) in at least 200 ml of water one time a day, approximately every 24 hours. (200 ml of water = 6.7 fluid ounces). Duration of study drug is 90 days. Participants in this arm of the study have different home medications prior to study enrollment than participants in the RCT treatment arm.
  Interventions: Drug: D-Mannose

INTERVENTIONS:
Drug: D-Mannose — A total of 2 g D-mannose daily
  Arms: Observational arm; RCT treatment arm

SUMMARY:
This is a study designed to evaluate the efficacy of a nutraceutical as a non-antibiotic treatment to prevent recurrent urinary tract infections in women that have completed menopause and are on vaginal estrogen therapy. An additional group of women with recurrent urinary tract infections that have completed menopause but are not using vaginal estrogen therapy will be followed while taking the nutraceutical. The study length is ninety days from the date that the study participant will be instructed is day 1.

DETAILED DESCRIPTION:
The objective of this study is to determine the efficacy of a nutraceutical as a non-antibiotic prophylaxis for postmenopausal women on vaginal estrogen therapy (VET) with a history of symptomatic, culture-proven recurrent urinary tract infection (rUTI) by means of a randomized, controlled trial. Recurrent urinary tract infections have a significant impact on patient health, quality of life, and finances (personal and societal).

The most common uropathogen for both acute and recurrent UTIs is Escherichia coli.

Historically, patients with rUTI have been placed on long-term prophylactic antibiotics to prevent recurrence. Long term antibiotic use can lead to antibiotic resistance, collateral damage to normal flora, and organ damage, such as pulmonary and hepatic toxicity with long-term nitrofurantoin use. There is an increasing prevalence of antibiotic resistance of uropathogenic E. coli and other uropathogens. Antibiotic resistance and its consequences have resulted in a need for non-antibiotic prophylaxis regimens.

A growing body of literature supports the use of vaginal estrogen therapy as a first-line non-antibiotic UTI prevention strategy in postmenopausal women. While VET has been shown to significantly reduce the risk of rUTIs, some women continue to have rUTIs. Other non-antibiotic strategies have been utilized including D-mannose, a nutraceutical. Three prior studies examined D-mannose as an isolated therapy with promising results, but in our experience, a multimodal approach has often been needed. Therefore, additional studies, such as this proposed research, are needed to determine the potential additive effect of a nutraceutical as a non-antibiotic prophylaxis for postmenopausal women using vaginal estrogen therapy.

ELIGIBILITY:
Inclusion Criteria:

For the RCT arms of the study, the following inclusion criteria will apply:

a. Postmenopausal women with recurrent UTI

i. Recurrent UTI defined as:

1. ≥ 2 symptomatic, culture-proven UTI in 6 months OR
2. ≥ 3 symptomatic, culture-proven UTI in 12 months

   ii. Postmenopausal defined as no menses for at least 12 months or surgical menopause

   b. At least one documented prior uropathogen susceptible to D-mannose

   c. Using VET for a minimum of four weeks prior to study day 1

   Inclusion criteria for the Observational arm of the study are the same with the exception of item 'c.' above (using VET for a minimum of four weeks) as participants will not be on vaginal estrogen therapy.

   Exclusion Criteria:

   For the RCT arms of the study, the exclusion criteria are as follows:
   1. Not postmenopausal
   2. Currently on daily antibiotic UTI prophylaxis (If this is the only exclusion criteria met, a woman could be cleared for inclusion in study/enrollment after a 2 week washout period occurs prior to inclusion in the study (RCT or Observational arm))
   3. Complicated UTIs (known renal tract anomaly, inability to empty bladder due to neurologic causes, performs self-catheterization or has an indwelling catheter)
   4. Patients with incomplete bladder emptying (defined as post void residual > 150 cc when minimal voided volume is >150 cc)
   5. Known contraindication to VET unless approved by patient's oncologist, oncologic surgeon, or primary care physician (History of or current endometrial cancer; History of estrogen sensitive breast cancer without approval of patient, patient's oncologist, oncologic surgeon, or primary care physician to use vaginal estrogen after counseling)
   6. History of interstitial cystitis/painful bladder syndrome
   7. Urothelial cancer
   8. Non-English speaking
   9. Enrolled in other clinical trials for UTIs
   10. Currently using D-mannose or Methenamine for UTI prevention

   Exclusion criteria for the Observational arm of the study are the same with the exception of item 'e.' above (known contraindication to VET) as participants will not be on vaginal estrogen therapy.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will involve only adult, postmenopausal women as recurrent UTI predominantly affect this population. Recurrent UTI in men would be considered complicated and would not be addressed with a prophylactic treatment like d-mannose.In addition, men do not go through menopause and do not have a vagina and would thus not be treated with vaginal estrogen therapy.
Enrollment: 61 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Lowder, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Derived] Lenger SM, Chu CM, Ghetti C, Durkin MJ, Jennings Z, Wan F, Sutcliffe S, Lowder JL. d-Mannose for Recurrent Urinary Tract Infection Prevention in Postmenopausal Women Using Vaginal Estrogen: A Randomized Controlled Trial. Urogynecology (Phila). 2023 Mar 1;29(3):367-377. doi: 10.1097/SPV.0000000000001270. Epub 2022 Oct 15. PMID 36808931
- [Derived] Lenger SM, Chu CM, Ghetti C, Durkin MJ, Jennings Z, Sutcliffe S, Lowder JL. Feasibility and Research Insights From a Randomized Controlled Trial for Recurrent Urinary Tract Infection Prevention in Postmenopausal Women Using Vaginal Estrogen Therapy. Female Pelvic Med Reconstr Surg. 2022 Jun 1;28(6):e163-e170. doi: 10.1097/SPV.0000000000001171. PMID 35421017

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 61 patients consented, 4 patients were in the observational arm and 57 were in the RCT arm (28 treatment, 29 control).
Period: Overall Study
Arm/Group | RCT Treatment Arm | RCT Control Arm | Observational Arm
Started | 28 | 29 | 4
Completed | 19 | 25 | 3
Not Completed | 9 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RCT Treatment Arm | RCT Control Arm | Observational Arm | Total
Number analyzed (Participants) | 28 | 29 | 4 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 13 | 1 | 23
  >=65 years | 19 | 16 | 3 | 38
Age, Continuous [Mean (Full Range); unit: years] | 70.7 [53 to 90] | 67.4 [50 to 83] | 71.5 [63 to 79] | 69.2 [50 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 4 | 61
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 28 | 4 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 26 | 28 | 4 | 58
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 4 | 61

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Symptomatic, Culture Proven Urinary Tract Infections
Description: To compare the cumulative incidence of symptomatic, culture-proven urinary tract infections in postmenopausal women with a history of rUTI on vaginal estrogen therapy randomized to receive prophylactic D-mannose versus women using vaginal estrogen therapy alone (control).
Time Frame: each participant will be followed for 90 days during study enrollment
Population: 57 patients were enrolled in the RCT(28 randomized to the treatment arm , 29 to the control arm). 4 participants in the Observational Arm. A total of 44 patients started study day1 across all three groups. Data was analyzed for 19 patients in the treatment arm and 25 patients in the control arm. Due to early termination and low recruitment in the Observational Arm, data on the 4 participants was not analyzed (1 withdrew prior to study day 1, 1 withdrew prior to completion - not study related).
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Treatment Arm | RCT Control Arm | Observational Arm
Number analyzed (Participants) | 19 | 25 | 2
Participants | 6 | 12 | 1

2. Secondary Outcome: Incidence of Symptomatic Culture Proved UTI From D-mannose Susceptible Uropathogens
Description: To compare the incidence of symptomatic, culture-proven urinary tract infections caused by all uropathogens potentially susceptible to D-mannose therapy in women receiving D-mannose and the control group. We will also compare these findings to the incidence of symptomatic, culture-proven urinary tract infections caused by uropathogens susceptible to D-mannose therapy in the absence of vaginal estrogen therapy (Control Arm).
Time Frame: each participant will be followed for 90 days during study enrollment
Population: There were 57 patients enrolled in the RCT (28 randomized to the treatment arm and 29 randomized to the control arm). There were 4 participants in the observational arm (data for 2 available for informal analysis; 1 withdrew prior to study day 1; 1 withdrew week 3 not related to study drug0. A total of 44 patients started study day 1 across all three groups. Data was analyzed for 19 patients in the treatment arm and 25 patients in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Treatment Arm | RCT Control Arm | Observational Arm
Number analyzed (Participants) | 19 | 25 | 2
Participants | 6 | 10 | 1

3. Secondary Outcome: Side Effects
Description: To describe the side effects of D-mannose and determine the incidence of discontinuation of therapy due to side effects.
Time Frame: each participant will be followed for 90 days during study enrollment
Population: There were 57 patients enrolled in the RCT (28 randomized to the treatment arm and 29 randomized to the control arm). There were 4 participants in the observational arm. A total of 44 patients started study day 1 across all three groups. Data was analyzed for 19 patients in the treatment arm and 25 patients in the control arm.
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Treatment Arm | RCT Control Arm | Observational Arm
Number analyzed (Participants) | 19 | 25 | 2
Participants | 3 | 0 | 0

4. Secondary Outcome: Incidence of Symptomatic, Culture Proven UTI in All Participants Taking D-mannose
Description: To compare the cumulative incidence of symptomatic, culture-proven urinary tract infections between women receiving prophylactic D-mannose treatment alongside vaginal estrogen therapy verses women receiving prophylactic D-mannose treatment whom are not on vaginal estrogen therapy (observational arm).
Time Frame: each participant will be followed for 90 days during study enrollment
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RCT Treatment Arm | RCT Control Arm | Observational Arm
Number analyzed (Participants) | 19 | 25 | 2
Participants | 6 | 12 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from dose day 1 through 90 days after treatment.
Arm/Group | RCT Treatment Arm | RCT Control Arm | Observational Arm
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29 | 0/4
Other Adverse Events (participants affected / at risk) | 14/27 | 16/29 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RCT Treatment Arm (N=27) | RCT Control Arm (N=29) | Observational Arm (N=4)
Flatulence (Gastrointestinal disorders) | 11 (15) | 5 (11) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (11) | 6 (15) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 5 (9) | 0 (0)

LIMITATIONS AND CAVEATS:
The primary limitation of this study was the low recruitment and retention encountered. Study retention was lower than expected. A futility analysis was performed at the interim analysis and we found that we do not have power to detect the effect size difference that we originally estimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03395288/Prot_SAP_007.pdf
  • Informed Consent Form (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT03395288/ICF_008.pdf